CLINICAL TRIAL: NCT01149798
Title: A Single Institutional Phase II Clinical Trial of Abraxane Combined With Cisplatin in Metastatic Breast Cancer
Brief Title: A Combination of Abraxane and Cisplatin in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Dr, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fudan BR2010-02
Record Dates: First submitted 2010-06-23; First posted 2010-06-24 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic breast cancer; combined chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Albumin-Bound Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abraxane and Cisplatin combination (Experimental): Abraxane and Cisplatin combination
  Interventions: Drug: Abraxane and Cisplatin combination

INTERVENTIONS:
Drug: Abraxane and Cisplatin combination — Abraxane will be given at 125 mg/m2, venous infusion within 30 minutes, administered on days 1, 8 and 15.
  Cisplatin at 75mg/m2, venous infusion for 120 minutes, will be administered on day 1.
  Other Names: Abraxane; Cisplatin

SUMMARY:
This phase II trial on the assumption that abraxane and cisplatin combination therapy is efficacy in metastatic breast cancer.

DETAILED DESCRIPTION:
The rationales for the combination of Abraxane and cisplatin include that either drug has antitumor activity; they have different mechanisms; no cross-resistance are documented between them, and there have been some preclinical evidences indicating synergistic effects between the two agents. This phase II study will be undertaken to evaluate combination of cisplatin and weekly abraxane in terms of efficacy and safety in MBC patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject must fulfill all of the following conditions or characteristics in order to be considered for study enrollment:

  1. Written informed consent prior to study specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time without prejudice.
  2. At least one measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST).
  3. Histopathologically or cytologically confirmed breast cancer.
  4. Female at an age of ≥18 years.
  5. Prior taxane or platinum treatment allowed. However, the drug interval should be longer than 12 months in adjuvant/neo-adjuvant setting and three months in MBC patients who have obtained ORR with taxane- or platinum-containing regimens.
  6. The lab values within 2 weeks prior to trial should meet:

     * PLT ≥100,000/mm3
     * ANC≥2000/mm3
     * HB≥80g/L
     * Total bilirubin < upper limit of normal level（UNL, < 1.5 x UNL for patients with liver metastasis)
     * ALT/AST < 1.5 x UNL (< 2.5 x UNL for patients with liver metastasis)
     * AKP < 5 x UNL (except for patients with bone metastasis)
     * Serum creatinine < UNL
  7. ECOG performance status of 0, 1 or 2.
  8. A life expectancy of more than 3 months.

Exclusion Criteria:

1. Pregnant or breast-feeding women.
2. Positive serum pregnancy test.
3. Unwilling to use a medically acceptable form of contraception, except for those who were surgically sterile or at least 1 year postmenopausal.
4. Uncontrolled brain metastases. Patients with brain metastases must be locally treated and the disease must be stable for at least one month at the time of enrolling.
5. Meningeal metastases.
6. Radiotherapy within the 4 weeks preceding study treatment start.
7. Incomplete recovery from the effects of major surgery.
8. Prior hormonal treatment allowed but must be discontinued 14 days prior to study entry.
9. Participation in any investigational drug study within 4 weeks preceding treatment start.
10. Blood transfusions or growth factors to aid hematological recovery within 2 weeks prior to study treatment start.
11. Significant medical condition that would make treatment or follow-up on this protocol difficult or problematic in the opinion of the treating oncologist.
12. Concurrent other malignancy at other sites or previous other cancer within the last 5 years, with the exception of adequately treated in situ carcinoma of cervix uteri or basal or squamous cell carcinoma of the skin or a contralateral breast cancer.
13. Serious uncontrolled intercurrent infections.
14. Poor compliance.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Overall response rates (ORR) of abraxane and cisplatin combination therapy | 2months

SECONDARY OUTCOMES:
Progression free Suivial (PFS) | 6 months
Number of adverse event | 2 months
Overrall Survival (OS) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, Study Chair — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China

REFERENCES:
- [Derived] Li Y, Zhao Y, Gong C, Xie Y, Hu X, Zhang J, Wang L, Zhang S, Cao J, Tao Z, Wang B. Cisplatin shows greater efficacy than gemcitabine when combined with nab-paclitaxel in metastatic triple-negative breast cancer. Sci Rep. 2019 Mar 5;9(1):3563. doi: 10.1038/s41598-019-39314-y. PMID 30837503
- [Derived] Tang LC, Wang BY, Sun S, Zhang J, Jia Z, Lu YH, Di GH, Shao ZM, Hu XC. Higher rate of skin rash in a phase II trial with weekly nanoparticle albumin-bound paclitaxel and cisplatin combination in Chinese breast cancer patients. BMC Cancer. 2013 May 9;13:232. doi: 10.1186/1471-2407-13-232. PMID 23659317